CLINICAL TRIAL: NCT03997838
Title: A Multicenter, Randomized, Double-Blind, Parallel Group, Placebo- Controlled Trial to Evaluate the Efficacy and Safety of VVZ-149 Injections for the Treatment of Post-Operative Pain Following Abdominoplasty
Brief Title: Evaluate the Efficacy and Safety of VVZ-149 Injections for the Treatment of Post-Operative Pain Following Abdominoplasty
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Vivozon, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: VVZ149-POP-P3-US003
Record Dates: First submitted 2019-05-28; First posted 2019-06-25 (Actual); Last update posted 2020-08-25 (Actual); Status verified 2020-08

CONDITIONS: Pain, Postoperative
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- VVZ-149 Injections (Experimental)
  Interventions: Drug: VVZ-149 Injections
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: VVZ-149 Injections — IV infusion of 1000 mg of VVZ-149
  Other Names: Opiranserin Injections
  Arms: VVZ-149 Injections
Drug: Placebo — IV infusion of 0 mg of VVZ-149
  Arms: Placebo

SUMMARY:
The purpose of this phase 3 study is to evaluate the efficacy and safety of an analgesic drug candidate, VVZ-149 Injections for treating post-operative pain following abdominoplasty.

ELIGIBILITY:
Inclusion Criteria:

* Men and women between 18-70 years old, inclusive. Female subjects must meet additional criteria according to childbearing potential.
* Planning to undergo abdominoplasty
* Ability to provide written informed consent
* Ability to understand study procedures and communicate clearly with the investigator and staff
* American Society of Anesthesiologists (ASA) risk class of I to II.

Exclusion Criteria:

* Emergency or unplanned surgery
* Previous abdominoplasty
* Pre-existing condition causing preoperative pain around the site of surgery
* Women who are pregnant or breastfeeding
* Chronic pain diagnosis and ongoing or frequent use of pain medications

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 307 (Actual)
Dates: Start 2019-05-23 (Actual); Primary Completion 2019-08-03 (Actual); Study Completion 2019-08-21 (Actual)

PRIMARY OUTCOMES:
Total Area Under the Curve (AUC) of Pain Intensity for 12 hours post-emergence | 0-12 hours post-emergence
  Using Numeric Pain Rating Scale (NRS, 0-10 at rest)

SECONDARY OUTCOMES:
Proportion of patients who report mild pain (NRS 0-3) at each time point during 24 hours post-emergence | 0-24 hours post-emergence
Total number of requests for rescue medication for 24 hours post-emergence | 0-24 hours post-emergence
Total amount of rescue medication consumption for 12 hours post-emergence | 0-12 hours post-emergence
Total amount of intra-operative fentanyl use | During surgery

CONTACTS AND LOCATIONS:
Overall Officials: Doo Lee, PhD, Study Chair — Vivozon, Inc.
Locations (5):
- United States (5):
  - Arizona Research Center, Phoenix, Arizona
  - Anaheim Clinical Trials, Anaheim, California
  - Midwest Clinical Research Center, Dayton, Ohio
  - Endeavor Clinical Trials, San Antonio, Texas
  - JBR Clinical Research, Salt Lake City, Utah

IPD SHARING:
Plan to Share IPD: No